CLINICAL TRIAL: NCT00889668
Title: Evaluation of the Performance and Use of GlucoTrack Model DF-F Non-Invasive Glucose Monitoring Device.
Brief Title: Evaluation of the Performance and Use of Non-Invasive Glucose Monitoring Device
Acronym: CR-01-001
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Integrity Applications Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CR-01-001 CTIL
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
Keywords: Glucose monitoring; GlucoTrack; Self glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): subjects with a diagnosis of type 1 or 2 diabetes; GlucoTrack results will be compared with the readings from approved invasive glucose meter device.
  Interventions: Device: GlucoTrack

INTERVENTIONS:
Device: GlucoTrack — comparison of different glucose monitoring devices

SUMMARY:
Diabetes is a leading cause of death in the Western World with medical costs increasing annually. There is no cure for diabetes, and blood glucose monitoring is a key component in diabetes treatment and management. Self-monitoring of blood glucose levels is essential to the self-management of diabetes and has become widespread over the past decade. Blood glucose determinations are currently done by invasive methods (finger tip pricking), followed by measuring the blood drop characteristics.

The purpose of this trail is to demonstrate the performance and use of GlucoTrack device in measuring blood glucose levels.

The rationale for development of the device is to improve the patient's quality of life by providing a device that is easily used and provides a painless measurement method, thereby leading to higher compliance, and to better managed diabetes

DETAILED DESCRIPTION:
See Brief summary

ELIGIBILITY:
Inclusion Criteria:

* Type 1or 2 Diabetes
* Anatomically suitable earlobe

Exclusion Criteria:

* Subjects requiring dialysis
* Any conditions that may hamper good contact between the PEC and the earlobe
* Pregnancy
* Nursing mothers

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2009-05; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Clarke Error Grid | one year

SECONDARY OUTCOMES:
User Satisfaction | one year
  Based on user questionnaire, user satisfection will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Harman-Boehm, MD, Principal Investigator — Soroka University Medical Center, Dept of Internal Medicine C and Director of the Diabetes Unit at Soroka University Medical Center
Locations (1):
- Soroka University Medical Center, Beersheba, Israel